CLINICAL TRIAL: NCT04474574
Title: How Differences in Oximeter Performance May Affect Clinical Decision: A Pragmatic Clinical Trial in Patients Under CPAP or Noninvasive Ventilation
Brief Title: How Differences in Oximeter Performance May Affect Clinical Decision
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Jean-Paul Janssens, Professor, University Hospital, Geneva
Other Study IDs: 2020-01813
Record Dates: First submitted 2020-07-13; First posted 2020-07-17 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Sleep Apnea; Alveolar Hypoventilation; Nocturnal Hypoxemia
MeSH Terms: conditions — Sleep Apnea Syndromes; Hypoventilation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Simultaneous recording of nocturnal SpO2 — The intervention will consist in performing a simultaneous recording of nocturnal SpO2 and pulse rate for at least 4 hours with 3 different devices.

SUMMARY:
In clinical practice discrepancies between overnight SpO2 recordings performed by 2 devices used simultaneously are regularly observed. However, this has not been systematically studied or quantified. It is therefore important to determine if these discrepancies are anecdotic, or frequent, and to what extent this may affect decisions in clinical practice such as implementing (or withdrawing) oxygen in subjects under noninvasive ventilation (NIV) or continuous positive airway pressure (CPAP), or adjusting NIV settings.

DETAILED DESCRIPTION:
Pulse oximetry estimates oxygen saturation in the arterial blood by trans-illuminating a translucent tissue (usually a fingertip, or an ear lobe) with light-emitting diodes at 2 specific wavelengths. Absorption of light at these different wavelengths (660 nm, red, and 940 nm, infrared respectively) differs between oxygenated and deoxygenated hemoglobin. The amount of light which is transmitted at both wave lengths is then quantified and processed by an algorithm that displays a saturation value. The signals are corrected for the pulsatile nature of arterial oxygen flow. Devices also provide pulse rate measured by plethysmography (pulse-related changes in volume of fingertip or earlobe). Since its introduction in the early 1980s, pulse oximetry has proven to be an essential tool for the non-invasive assessment of blood oxygen saturation (SpO2). The use of pulse oximeter is now widespread and interests acute care settings as well as primary care settings. Although there have been recent improvements in signal analysis such as increasing sampling frequency and improving reflectance technology [4], the accuracy of commercially available oximeters differs. First of all, there is variability in the way accuracy of pulse oximetry devices is reported within 2% (± 1 SD) or within 5% (± 2 SD) of reference measurements obtained by blood gases analysis [5]. Secondly, there is a variability between commercially available devices, especially below a SpO2 of 90%. This is partly explained by the fact that calibration of the different algorithms employed in signal processing is limited by the range of saturations that can be safely obtained in healthy volunteers. In respiratory medicine, it has been shown that such variability of accuracy could affect the diagnosis of Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS) and impact on clinical decisions as the recorded number of apneas/hypopneas varied between devices during nocturnal sleep studies [8] Nocturnal hypoxemia (NH) is considered as one of the major determinants of adverse cardiovascular complications and neurocognitive impairment in patients suffering of chronic respiratory failure (CRF). Because of its simplicity, short set-up time and short time response, pulse oximetry is a valuable screening tool for nocturnal hypoxemia despite its disadvantages such as motion artefacts or sensitivity to perfusion. Therefore, definitions of NH rely solely on nocturnal oximetry recording: for instance, in a consensus statement on noninvasive ventilation, spending > 5% of sleep time under 88% of SpO2 was considered as a relevant threshold. Definitions of NH remain arbitrary and different expert-based thresholds have been suggested in the medical literature [10]. Patients suffering from nocturnal hypoventilation, especially those with an average daytime SpO2 close to the steep portion of the hemoglobin dissociation curve (SpO2 between 90-94%), are at higher risk for NH. Therefore, in these patients, device imprecision could have a significant impact on medical decisions, such as deciding to adjust ventilator settings in patients under noninvasive ventilation (NIV) and/or implementing nocturnal oxygen supplementation.

In patients with CRF and NIV, after optimal adjustment of ventilator settings, prescription of nocturnal oxygen supplementation is common practice although impact of nocturnal oxygen supplementation on survival, patient comfort, or prevention of cor pulmonale has yet to be demonstrated. Practically speaking, it increases considerably the burden of the treatment for the patient and care givers (additional connections and tubings, noise of the oxygen concentrator etc.). To our knowledge, no study has evaluated how the use of different pulse oximeters could impact on this decision. Three types of devices are used in clinical practice: pulse oximetry using a probe connected to the home ventilator device, pulse oximetry combined with transcutaneous capnography, or using a "wrist watch" type of device.

ELIGIBILITY:
* Inclusion criteria:

  * > 18 years old
  * Awake room air SpO2 between 90 and 94%
  * NIV or CPAP therapy
  * Ambulatory or hospitalized patient in a clinically stable respiratory condition without any vasopressor treatment.
* Exclusion criteria:

  * Hospitalization in an acute care setting (e.g. emergency room, Intensive Care Unit, Intermediate Care Unit)
  * Any vasopressor treatment
  * Peripheral vascular pathologies that can affect digital perfusion (e.g. history of ischemia, Raynaud's phenomenon, any type of vasculitis).
  * Mechanical obstacles that may limit quality of signal (e.g. nail polish, bandage, splint, plaster).
  * Patient already treated by long term nocturnal oxygen therapy (LTOT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited among 1) hospitalized patients with NIV treatment; 2) ambulatory patients followed for NIV therapy at the outpatient unit of the Division of Pulmonology; 3) patients undergoing an elective polysomnography (sleep study) for adjustment or titration of a positive pressure device (NIV or CPAP) at the Sleep Laboratory of the Division of Pulmonology.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Degree of agreement | 3 months
  The primary endpoint is the degree of agreement between 3 different devices used simultaneously for overnight SpO2 recording for 3 commonly used threshold values defining nocturnal hypoxemia: 5% of time with an SpO2 < 88%, 10% of time with an SpO2 < 90% or 20% of time with an SpO2 < 90%.

SECONDARY OUTCOMES:
Bland and Altman analysis of agreement | 3 months
  Bland and Altman analysis of agreement between devices , two by two (A vs B, A vs C)
Degree of agreement with threshold values | 3 months
  an analysis of agreement of oxygen desaturation index between devices, comparing devices 2 x 2, and using a threshold value of 10/hour as clinically significant
Minimal SpO2 value | 3 months
  a comparison of the minimal SpO2 value and time spent under different threshold levels (88 and 90%) between devices
Mean pulse rate | 3 months
  A comparison of average pulse rate between devices

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Karege G, Egger B, Lawi D, Bergeron A, Janssens JP. How Using Different Oximeters May Affect Clinical Decision-Making: A Method Comparison Study in Patients Receiving CPAP or Noninvasive Ventilation. Chest. 2026 Jan;169(1):244-256. doi: 10.1016/j.chest.2025.08.018. Epub 2025 Sep 9. PMID 40930342